CLINICAL TRIAL: NCT00212719
Title: Controlled Study of ONO-5920 in Patients With Involutional Osteoporosis in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-5920-03
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Involutional Osteoporosis
Keywords: ONO-5920, osteoporosis, bisphosphonate
MeSH Terms: conditions — Osteoporosis | interventions — YM 529

INTERVENTIONS:
Drug: ONO-5920

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ONO-5920 in patients with involutional osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis in accordance with Criteria for the Diagnosis of Primary Osteoporosis.
2. Other inclusion criteria as specified in the study protocol.

Exclusion Criteria:

1. Patients having secondary osteoporosis or another condition that presents low bone mass.
2. Patients having findings that affect measurement of lumbar spinal bone mineral density by DXA
3. Patients that have been administered bisphosphonate derivatives.
4. Other exclusion criteria as specified in the study protocol.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2003-05; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Mean bone mineral density of the lumbar spine (L2-4 BMD)

SECONDARY OUTCOMES:
Bone mineral density at femur, fragility fractures, biochemical markers of bone turnover, lower back pain

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, ' Development Planning, Study Director — Ono Pharmaceutical Co. Ltd

REFERENCES:
- [Derived] Hagino H, Nishizawa Y, Sone T, Morii H, Taketani Y, Nakamura T, Itabashi A, Mizunuma H, Ohashi Y, Shiraki M, Minamide T, Matsumoto T. A double-blinded head-to-head trial of minodronate and alendronate in women with postmenopausal osteoporosis. Bone. 2009 Jun;44(6):1078-84. doi: 10.1016/j.bone.2009.02.016. Epub 2009 Mar 2. PMID 19264155